CLINICAL TRIAL: NCT00534326
Title: Standard Reaming Versus Reaming/Irrigating/Aspirating for Intramedullary Nailing of Femoral Shaft Fractures
Acronym: STAFF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prisma Health-Upstate (Other)
Collaborators: University of Missouri-Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Ort-07-06-06
Record Dates: First submitted 2007-09-20; First posted 2007-09-24 (Estimated); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Femoral Fractures
MeSH Terms: conditions — Femoral Fractures

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Standard Reaming of femoral shaft fracture prior to intramedullary nailing
  Interventions: Procedure: Standard Reaming
- 2 (Active Comparator): Reamer/Irrigator/Aspirating of femoral shaft fracture prior to intramedullary nailing
  Interventions: Procedure: Reaming/Irrigating/Aspirating

INTERVENTIONS:
Procedure: Standard Reaming — Femoral reaming using standard reaming techniques of multiple reamers
  Arms: 1
Procedure: Reaming/Irrigating/Aspirating — Reaming using the Reamer/Irrigator/Aspirating
  Arms: 2

SUMMARY:
Reaming (enlarging of the bone canal) is commonly performed prior to the insertion of intramedullary nails for the fixation of long bone fractures. This study is designed to compare the union rates between fractures reamed by standard reaming versus reaming with a Reamer/Irrigator/ Aspirator (RIA). In addition, this study will collect patient-based outcomes on these patients. Little information exists on the patient based outcomes following femur fractures. We hope that the patient based outcomes of this study will also be able to aid physicians in advising patients with femur fractures of their possible outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women between the ages of 18 years and 85 years;
2. Acute fractures of the femoral shaft

Exclusion Criteria:

1. Fractures not amenable to intramedullary nailing and deemed by the treating surgeon;
2. Pathological fractures;
3. Open fractures;
4. Patients with additional injuries to the ipsilateral femur;
5. Surgical delay of greater than 7 days from the time of injury;
6. Retained hardware in the affected limb;
7. Previous infection in fractured limb;
8. Likely problems in the judgment of the investigators with maintaining follow-up;
9. Patients with severe cognitive injuries or disabilities will be excluded if it is deemed that they will be unable to complete the study questionnaires;
10. Hopeless diagnosis;
11. Medical comorbidities that prohibit the conductance of surgical treatment under a general anesthetic;
12. Fractures requiring cephalomedullary nails

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2006-12; Primary Completion 2015-12 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
Fracture Healing | 3 months, 6 months, 1 year, 2 years

SECONDARY OUTCOMES:
Patient Based Quality of Life | Baseline, 3 months, 6 months, 1 year, 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Kyle J Jeray, MD, Principal Investigator — Prisma Health-Upstate
Locations (9):
- United States (9):
  - Indiana University, Indianapolis, Indiana
  - Lahey Clinic, Burlington, Massachusetts
  - University of Missouri- Columbia, Columbia, Missouri
  - Carolinas Medical Center, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Palmetto Health, Columbia, South Carolina
  - Greenville Hospital System Univeristy Medical Center, Greenville, South Carolina
  - University of Tennessee-Chattanooga Unit, Chattanooga, Tennessee
  - Carilion Medical Center, Roanoke, Virginia